CLINICAL TRIAL: NCT02946762
Title: Z 31501 - Treatment as Prevention (TasP) in Correctional Facilities in Zambia and South Africa
Brief Title: TasP in Correctional Facilities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Department for International Development, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 15-1473
Record Dates: First submitted 2016-09-14; First posted 2016-10-27 (Estimated); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: HIV; Tuberculosis
Keywords: HIV; TB; Antiretroviral Treatment; Anti-tuberculosis Treatment; HIV Counselling and Testing; Treatment as Prevention
MeSH Terms: conditions — Tuberculosis | interventions — Coal Tar

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Universal Test and Treat (Other): All incarcerated individuals with HIV infection will receive antiretroviral therapy (ART) by test and treat.
  Interventions: Other: Test and treat

INTERVENTIONS:
Other: Test and treat — All incarcerated individuals found to have HIV infection will be offered universal voluntary HIV counseling and testing (HCV) through routine care provided at the correctional facility followed by referral to the study for immediate (routine, non-study prescribed) ART, regardless of CD4 cell count. The ART regimen prescribed will be the standard first-line, fixed-dose combination efavirenz plus lamivudine/emtricitabine and tenofovir per Zambian national guidelines.

SUMMARY:
At correctional facilities in Zambia and South Africa, a cross-sectional study design will be used to characterize the full continuum of integrated HIV/TB care under Treatment as Prevention (TasP), and will enrich this approach by: 1) using individual-level cohort data for HIV-infected inmates to assess ART uptake under TasP/Universal Test and Treat (UTT), as well as 6-month virological suppression and retention in care for inmates initiating ART; and 2) mixed methods to identify health-system, corrections-related socio-cultural and individual-inmate barriers to and facilitators of TasP/UTT to refine TasP implementation; and 3) conducting a retrospective chart review using routine data from Ministry of Health registers to reconstruct an approximate HIV and TB cascade for all inmates (HIV-infected and HIV-uninfected) at 3 and 12 months into TasP/UTT implementation.

DETAILED DESCRIPTION:
Treatment as Prevention (TasP) offers promise to: (1) prevent HIV transmission among incarcerated populations; and (2) improve inmate health and tuberculosis control through provision of immediate ART using a "universal test and treat" (UTT) approach.

Increased uptake of routine HIV counseling and testing (HCT) services will be encouraged and currently available ART care will be augmented by offering immediate ART initiation to all HIV-infected inmates not already on ART (after screening for TB and kidney disease) regardless of CD4 count. In this way, the study will promote universal HCT and ART access.

Existing, routine service delivery platforms operated by the MOH and Zambia

Corrections Service will be strengthened in hopes of achieving the following:

1. Universal HIV testing within 2 months of facility entry and annually for all current inmates
2. Clear integration of TB screening and treatment within HIV care services
3. Scaling-up inmate peer supporters and support groups to promote ART adherence
4. Strengthened systems for providing integrated TB/HIV care in correctional settings
5. Improved continuity of care for prisoners initiating ART

The following study-specific procedures will be carried out:

* ART will be initiated following clinical and laboratory assessment according to local guidelines.
* All inmates with newly diagnosed or previously documented HIV infection will be offered immediate ART regardless of CD4+ count or WHO clinical stage. A clinical assessment, including TB screening, and testing of serum creatinine will be completed, per Zambian national guidelines, prior to starting a standard ART regimen, which in Zambia is efavirenz plus lamivudine/ emtricitabine and tenofovir.
* A study specific follow-up visit, aligned with the routine HIV care schedule, for all inmates identified as HIV-infected will occur:
* Study nurses will support blood sample collection for HIV-1 viral load monitoring at the single study follow-up visit for all participants initiating ART under TasP. The planned follow-up visit will be scheduled to occur at 6 months following ART initiation. However, if a high recidivism rate and loss to follow-up prior to 6 months on treatment is observed, the study follow-up visit may be moved up to 3 months.

Study data collection will augment existing routine data collection mechanisms and allow individual-level outcome ascertainment regarding uptake of ART under TasP, as well as 6-month retention in care and virological suppression.

Standardized questionnaires and in-depth interviews will be conducted with inmate participants enrolled under Objective 1. To assess systems-level issues, in-depth interviews will also be conducted with a purposive sample of correctional staff and health care workers.

ELIGIBILITY:
Inclusion Criteria:

* Previously known or newly diagnosed HIV-infected inmates
* Not on ART
* No documented release date within 30 days of enrollment
* Incarcerated in an adult correctional ward at one of the three study sites.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 419 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
Proportion of inmates with HIV-infection who were assessed for and offered ART initiation under TasP/UTT | 2 years

SECONDARY OUTCOMES:
Proportion of all HIV-infected inmates starting ART who are retained on ART among those who remain in the study facility | 2 years
Proportion of inmates on ART with an HIV RNA <40 c/mL at 6 months of ART | 6 months
Proportion of HIV-infected inmates with TB diagnosis who initiate anti-TB therapy under TasP/UTT | 2 years
Proportion of inmates on ART with an HIV RNA <40 c/mL at 12 months of ART | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael Herce, MD, MPH, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Lusaka Central Corrections ART Clinic, Lusaka, Zambia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Herce ME, Hoffmann CJ, Fielding K, Topp SM, Hausler H, Chimoyi L, Smith HJ, Chetty-Makkan CM, Mukora R, Tlali M, Olivier AJ, Muyoyeta M, Reid SE, Charalambous S. Universal test-and-treat in Zambian and South African correctional facilities: a multisite prospective cohort study. Lancet HIV. 2020 Dec;7(12):e807-e816. doi: 10.1016/S2352-3018(20)30188-0. Epub 2020 Aug 4. PMID 32763152